CLINICAL TRIAL: NCT06717399
Title: Pilot Study: The Effects of Telehealth Mindfulness Meditation Program on Sleep Quality and Anxiety in Acquired Brain Injury Population
Brief Title: Effect of Telehealth Mindfulness on Sleep and Anxiety in Acquired Brain Injury Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Joseph's University, Philadelphia (Other)
Responsible Party: Principal Investigator, Nabila Enam, Clinical Associate Professor, Saint Joseph's University, Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StJosephU
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Acquired Brain Injury
Keywords: Sleep; Anxiety; mindfulness meditation; Acquired brain injury
MeSH Terms: conditions — Brain Injuries; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, one-group pretest-posttest, quantitative design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eight- session of mindfulness meditation (Experimental): Each mindfulness meditation session will be 30 minutes long, consisting of a 5-minute introduction, 15 minutes of guided mindfulness meditation, and 10 minutes of educational discussion. Participants are required to complete two mindfulness meditation sessions per week. Participants must complete a minimum of 8 sessions over 4 to 5 weeks.
  Interventions: Other: Mindfulness meditation

INTERVENTIONS:
Other: Mindfulness meditation — Each mindfulness meditation session will be 30 minutes long, consisting of a 5-minute introduction, 15 minutes of guided mindfulness meditation, and 10 minutes of educational discussion.

SUMMARY:
The goal of this study is to learn the effect of a telehealth mindfulness meditation program on sleep quality and anxiety in individuals with brain injury living in the community. The main questions it aims to answer are:

* Does an eight-session mindfulness meditation program change sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) in individuals with acquired brain injury?
* Does an eight-session mindfulness meditation program change anxiety levels as assessed by the Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form in individuals with acquired brain injury?

Participants will:

* Complete eight sessions of mindfulness meditation over 4 to 5 weeks
* Complete two mindfulness meditation sessions per week.
* Complete two additional sessions for pre- and post-test measurements.

DETAILED DESCRIPTION:
This is a pilot study examining the effects of a mindfulness meditation program on sleep quality and anxiety levels in individuals with acquired brain injury living in the community. Participants will receive a thirty-minute mindfulness meditation session. Each thirty-minute session will consist of five minutes of introduction, 15 minutes of guided mindfulness meditation, and 10 minutes of education and discussion. Participants will need to complete eight sessions of mindfulness meditation and pre-and post-tests to be included in the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of acquired brain injury
* Score 19 or below on the Short Orientation-Memory-Concentration Test of Cognitive Impairment (SOMC)
* 18 years or older
* Can speak and comprehend English
* Have access to an internet connection and an electronic device

Exclusion Criteria:

• Diagnosis of aphasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Associate Professor, OTD, Principal Investigator — Saint Joseph's University
Locations (1):
- Saint Jospeh's University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available by the primary investigator upon request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was rolling, starting after IRB approval (January 6, 2025), and the last recruitment day was February 28, 2025. The study utilized convenience, non-probability sampling in which emails and flyers were sent and posted in the community through ABI support groups and associations such as the Pennsylvania Brain Injury Association, the Brain Injury Alliance of New Jersey, the Brain Injury Association of Delaware, SJU campuses, and word of mouth.
Pre-assignment Details: Participants were only included in the study if they met the inclusion criteria. They were eligible for this study if they had a known diagnosis of acquired brain injury, scored 19 or below on the SOMCT, were 18 years or older, could speak and comprehend English, and had access to an internet connection and an electronic device. Participants were excluded from the study if they had a diagnosis of aphasia.
Groups:
- Eight- Session of Mindfulness Meditation: Each mindfulness meditation session was 30 minutes long, consisting of a 5-minute introduction, 15 minutes of guided mindfulness meditation, and 10 minutes of educational discussion. Participants were required to complete two mindfulness meditation sessions per week. Participants must complete a minimum of 8 sessions over 4 to 5 weeks.
Period: Overall Study
Arm/Group | Eight- Session of Mindfulness Meditation
Started | 12
Completed | 11
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eight- Session of Mindfulness Meditation
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.91 (16.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
the Pittsburgh Sleep Quality Index (PSQI) and PROMIS Anxiety Short Form [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report tool assessing sleep quality over the past month. It includes seven components scored from 0-3, with a global score ranging from 0-21. A score >5 indicates poor sleep quality. The The Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form is an 8-item measure assessing anxiety over the past 7 days using a 5-point Likert scale (1-5). Total scores range from 8-40, with higher scores indicating greater anxiety.
  units on a scale
    PSQI | 7.73 (3.17)
    PROMIS Anxiety Short Form | 58.18 (4.30)

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburg Sleep Quality Index assesses sleep disturbances and quality through a self-rated questionnaire. The 19-question self-reported assessment has seven subcategories. The questionnaire is made up of scaled responses from 0-3; 0 is not during the past month, 1 is less than once a week, 2 is once or twice a week, and 3 is three or more times a week. The minimum total score is 0, maximum score is 21.If the individual scores higher than a 5 overall, it is an indication of poor sleep quality.
Time Frame: Pre-test Before the start of the intervention (baseline) and Post test after the completion of 8 sessions of mindfulness meditation, up to 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eight- Session of Mindfulness Meditation
Number analyzed (Participants) | 11
units on a scale
  Pre- test | 7.73 (3.17)
  Post -test | 4.00 (2.66)
Statistical Analysis 1: Comparison: Eight- Session of Mindfulness Meditation; Null Hypothesis: ● There will not be a change in sleep quality after participation in eight mindfulness meditation sessions as measured by the Pittsburgh Sleep Quality Index; Test type: Other — The number of participants (n=15) was calculated using an effect size of 0.89. This effect size was based on a randomized clinical trial utilizing a structured mindfulness meditation program on moderate sleep disturbances in older adults (Black et al. 2015). A power of 0.8 and a significance level of 0.05 was utilized to calculate the sample size, a minimum of 12 participants is required to demonstrate significance in this study. To account for 20% attrition total participants needed is 15; p = 0.00058, t-test, 2 sided

2. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form
Description: The Patient Reported Outcomes Measurement Information System Anxiety Short Form is an eight-question self-report measure to assess anxiety. Participants will be asked to rate their responses to questions relating to feelings of anxiety in the past seven days. Participants will rate their feelings using a 5-point Likert scale, where answers can range from 1-5. One corresponds with "never," 2 with "rarely," 3 with "sometimes," 4 with "often," and 5 with "always." Lowest possible raw score is 8, and the highest possible raw score is 40. Raw scores are converted into T-scores. T-scores conversion ranges from 30 to 80. The higher score indicates a greater severity of anxiety. The general population mean for T-score is 50, and the Standard deviation is 10. A T-score of less than or equal to 55 is indicative of within normal limits, T-scores between 55- 60 mild, a score between 60-70 moderate, and a score > 70 severe anxiety.
Time Frame: Pre-test Before the start of the intervention (baseline) and Post-test after the completion of 8 sessions of mindfulness meditation, up to 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eight- Session of Mindfulness Meditation
Number analyzed (Participants) | 11
units on a scale
  Pre-test | 58.18 (4.30)
  Post-test | 52.99 (3.82)
Statistical Analysis 1: Comparison: Eight- Session of Mindfulness Meditation; Test type: Other; p = 0.004, t-test, 2 sided

3. Other Pre Specified Outcome: Patient Global Impression of Change (PGIC)
Description: The Patient Global Impression of Change is one question in a Likert-scale form for the participants to provide feedback about how the program ran. The scale ranges from 0 to 6. 0 corresponds with "very much improved," 1 with "much improved," 2 with "minimally improved," 3 with "no change," 4 with "minimally worse," 5 with "much worse," and 6 with "very much worse." The minimum score possible on the measurement is 0, and the maximum score possible is 6. The lower score on the measurement indicates improvement.
Time Frame: Post- test After the completion of 8 sessions of mindfulness meditation, up to 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eight- Session of Mindfulness Meditation
Number analyzed (Participants) | 11
units on a scale | 2.36 (0.50)

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: The subject's death was due to a medical condition and not related to the study.
Arm/Group | Eight- Session of Mindfulness Meditation
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
The study may have had attentional bias due to participants' heightened awareness of their sleep quality and anxiety when completing self-reported outcome measures. Additional limitations are non-probability convenience sampling as a recruitment method. This method of recruitment does not provide an accurate representation of the ABI population. The positive outcomes cannot be attributed to the mindfulness meditation sessions alone, due to the lack of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT06717399/Prot_SAP_000.pdf